CLINICAL TRIAL: NCT05122611
Title: Post Lumbar Radiofrequency Neurotomy Imaging
Status: Completed | Type: Observational
Sponsor: FUSMobile Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RFMRI01
Record Dates: First submitted 2021-08-20; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-08

CONDITIONS: Facet Joint Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention, imaging study only — Imaging study only

SUMMARY:
MRI imaging post radio frequency ablation procedure for facet arthritis

DETAILED DESCRIPTION:
This study is an imaging study. Following a radio frequency ablation procedure for facet arthritis low back pain the patient can join the imaging study.

During the study the patient undergo contrast enhanced MRI imaging of the lumbar spine Once the imaging is done the patient finishes the study

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and females, legally able and willing to participate in the study
2. Able and willing to complete the research questionnaires and communicate with the investigator and research team
3. Patients who are scheduled to have bilateral or unilateral treatment by radiofrequency neurotomy for chronic lumbar pain.

Exclusion Criteria:

1. Pregnant or breastfeeding patient
2. Patients younger than 18
3. Patients unable to understand and complete the research questionnaires in English
4. Patient with any contraindication for MRI contrast agents - Patients with known intolerance or allergies to the MRI contrast agent (e.g., Gadovist) including advanced kidney disease
5. Patients with a pacemaker, implanted defibrillator or internal pacing wires.
6. Patient with mechanical heart valve
7. Patient with an aneurysm clip
8. Patient with eye surgery or injury involving a metallic object
9. Patient with ear surgery or implanted device to the ear
10. Patient with any implanted electrical, metallic or magnetic device such as implanted neurostimulator, implanted drug infusion pump or bone growth stimulator
11. Patient with any kind of prosthesis (Eye, Ear, Penile, limb), or any other metal in your body from surgery or injury
12. Patient with vascular clamp, filter, coil or stent
13. Pregnant or breast-feeding patient
14. Patient with anemia, liver disease or history of MRI contrast reaction
15. Patient with any known kidney disease, prior kidney surgery or on dialysis
16. Patient with hypertension or diabetes that requires medication
17. Patient with any metal in or on their body (example: shrapnel, BB's, Tattoos, permanent makeup)
18. Patients who are claustrophobic or known adverse psychological reactions with previous MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients volunteering to receive an MRI scan with and without contrast following radiofrequency neurotomy treatment for chronic lumbar pain
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
MRI imaging of the lumbar spine | Up to 5 days after the RFA procedure (which was done before the study)
  MRI imaging of the lumbar spine

CONTACTS AND LOCATIONS:
Locations (1):
- Silver Medical Group, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No